CLINICAL TRIAL: NCT04477161
Title: Effect of Ketone Esters on Parkinson Disease: A Pilot, Prospective Trial.
Brief Title: Effect of Ketone Esters in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Ketone in PD; IRB201901326 (Other: UF IRB); OCR24402 (Other: UF OnCore)
Record Dates: First submitted 2020-06-22; First posted 2020-07-20 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Parkinson Disease; Ketosis
Keywords: parkinson disease; ketosis; microbiota
MeSH Terms: conditions — Parkinson Disease; Ketosis

STUDY DESIGN:
Intervention Model Description: pilot, prospective, single-arm, single-center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketone Intervention (Experimental): Subjects will take the Ketone Ester Elite Endurance Nutrition Drink. They will drink 1 bottle 4 times daily for 4 weeks
  Interventions: Dietary Supplement: Ketone Ester Elite endurance Nutrition Drink; Other: Stool Sample

INTERVENTIONS:
Dietary Supplement: Ketone Ester Elite endurance Nutrition Drink — Subjects will take one bottle four times daily for four weeks
Other: Stool Sample — Subjects will provide a stool sample at 2 timepoints.

SUMMARY:
Ketones esters have shown to improve mitochondrial function and are currently use to enhanced functional performance. As Mitochondrial dysfunction is one of the proposed mechanism of neuronal injury in Parkinson's disease, the study aims to assess the tolerability,side effects and effect of oral ketone esters in Patients with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a debilitating progressive neurodegenerative disorder, second in frequency only to Alzheimer's disease, affecting around 10 million people worldwide. PD is characterized by loss of dopaminergic cells in substantia nigra and the accumulation of Lewy bodies. There is no disease modifying treatment or cure for the disease and management strategies focus on symptomatic treatment. One of the proposed mechanisms for the dopaminergic neurons degeneration in sporadic Parkinson's disease cases is related to compromise cellular bioenergetics, resulting in excessive production of reactive oxygen species (ROS) that leads to oxidative stress. Numerous studies have identified mitochondrial dysfunction as the central pathological features of both genetic and sporadic PD. Mitochondrial dysfunction can also increase inflammation which is associated with PD and Lewy Body formation. Elevated plasma ketones have been shown to enhance energy reserves, ATP levels and the expression of many enzymes involved in multiple metabolic pathways in the mitochondria. This pilot study aims to assess the effect of an exogenous ketone supplement on functional performance in people with PD. Changes in inflammatory makers will also be assessed. Participants will ingest the exogenous ketone supplement four times per day for four weeks. Participants will undergo neurological, functional, and cognitive assessments prior to and after the four-week intervention. Dietitians will follow up with participants weekly for compliance and counseling. Diet will be assessed throughout the study using the automated self-administered 24-hour dietary recall. After the four week intervention, a two-week "washout" period will be observed before reassessing functional and cognitive performance again.

Additionally, the study would like to establish the extent to which the use of Ketone esters impact the gut microbiota. Gut microbita composition in PD has been associated with symptoms and treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed Parkinson's Disease
* 40-75 years of age
* On stable dopaminergic therapy
* Willing and able to complete the informed consent form in English
* Willing to consume the study supplement four times each day during the 4-week intervention period
* Willing to complete all dietary recalls over approximately 6 weeks
* Willing to complete all daily and weekly questionnaires throughout the six weeks.

Exclusion Criteria:

* Does not meet the above criteria
* Atypical or secondary Parkinsonism
* BMI >30
* Rheumatological or other inflammatory conditions
* Following of the ketogenic diet
* History of ulcer disease
* History of irritable bowel disorder or irritable bowel syndrome
* Currently taking any medication that could affect stool formation.
* Diagnosis of Diabetes mellitus Type 1 or Type 2
* Currently smoking (including vaping) tobacco products.
* Women who are lactating, know that they are pregnant, or are attempting to get pregnant.
* Note: a pregnancy test will be administered prior to initiating consumption of the study supplement. Women who are pregnant will be withdrawn from the study at that time.
* Use of another investigational product within 3 months of the initial visit.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Changes in serum Ketones | Baseline up to 4 months
  by measuring the beta-hydroxybutyrate/serum glucose levels in blood at baseline and four months

CONTACTS AND LOCATIONS:
Locations (1):
- Fixel Institute for Neurological Diseases, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will be shared with collaborators on project here at the University of Florida and only de-identified data will be released with IRB approval.